CLINICAL TRIAL: NCT00823641
Title: An Open, Non-randomised Pilot Study of Anti-TNF-alpha Therapy in Early or Progressing HAM/TSP
Brief Title: The HAM Infliximab Study
Acronym: HAM06
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Higher toxicity rate than observed in studies in Rheumatoid arthritis
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Graham Taylor, Reader in Communicable Diseases, Imperial College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cro948; EUDRACT: 2007-005554-23
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: HTLV-I-associated Myelopathy
Keywords: HAM/TSP; HTLV-I
MeSH Terms: conditions — Paraparesis, Tropical Spastic | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infliximab (Experimental): Infliximab 3mg/kg infused intravenously at weeks 0, 2 and 8 and then every 8 weeks until and including week 40 of the study
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab 3mg/kg infused intravenously at weeks 0, 2 and 8 and then every 8 weeks until and including week 40 of the study

SUMMARY:
An open-label, non-randomised, uncontrolled, proof-of-concept study of eight patients with 'definite' HTLV-I-associated myelopathy/Tropical Spastic Paraparesis (HAM/TSP). Eligible patients will have either early disease (of less than 2 years duration) or progressive disease (with observed clinical deterioration during the preceding 3 months.

Following 2 baseline assessments including Magnetic Resonance Imaging (MRI) of the spinal cord and a lumbar puncture for examination of the fluid around the brain (CSF) participants will be treated with a total of 7 infusions of the anti-TNF-alpha antibody infliximab over a period of 48 weeks. After the last on therapy assessment at 48 weeks participants will be followed up for a further 24 weeks. Study assessments will be clinical, virological, immunological and radiological. MRIs of the spinal cord will be obtained at weeks 12 and 72. CSF will be examined, on therapy, at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Are able to give informed consent
* Are 16 years or older
* Have 'definite' HAM/TSP according to the criteria of "Definite HAM/TSP" agreed in Belem 200361
* Have early or progressing disease as defined here:

  * "Early HAM/TSP": Patients must have motor disability (minimum of stiffness or weakness) for less than 2 years. (Bladder symptoms if the original and only presenting symptoms as assessed by history are not included)
* "Progressing HAM/TSP"
* New or worsening motor symptoms in a patient with definite HAM of > 2 years duration within the last 3 months

Exclusion Criteria:

* Hepatitis B or hepatitis C infection
* HIV infection
* Overt sepsis, abscesses or opportunistic infections
* Active TB (untreated or on treatment)
* Strongyloides stercoralis (untreated)
* Known hypersensitivity to inflixmab, other murine proteins or to any of the excipients
* Malignancy
* Moderate or severe heart failure (NYHA class III/IV)
* Pregnancy or breastfeeding
* Unhealed surgical wounds
* Planned impending surgery - treatment would be withheld for 2-4 weeks prior to major surgery and started/restarted post-operatively if no evidence of infection and wound healing is satisfactory
* Current immunosuppressive or immunomodulatory therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical failure | 48 weeks

SECONDARY OUTCOMES:
Change in timed 10m walk | 12, 24, 48 and 72 weeks
Clinical Safety | 48 weeks
HTLV-I viral load in CSF | 12 weeks
HTLV-I viral load in peripheral blood | 12, 24, 48 and 72 weeks
% CD4+ T- lymphocytes expressing CD25 | 24, 48 and 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Graham P Taylor, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom